CLINICAL TRIAL: NCT04113707
Title: Building Long-term Academic Success Through Ongoing Fun Fitness Program
Acronym: BLASTOFF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI has left the institution
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-0180
Record Dates: First submitted 2019-09-30; First posted 2019-10-03 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Reading Disorder
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Intervention Model Description: Pre and post two group intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Lab (Experimental): Group A will receive 20 minutes of motor lab intervention daily.
  Interventions: Behavioral: Motor lab activity
- Standard of Care (No Intervention): Group B will receive standard of care which will be 20 minutes of reading per day.

INTERVENTIONS:
Behavioral: Motor lab activity — fitness, gross motor, fine motor, and motor coordination activities
  Arms: Motor Lab

SUMMARY:
The purpose of the research study is to investigate if daily motor activities, including fitness activities, gross motor skills, fine motor skills, and motor coordination activities result in physiological, cognitive, and behavioral benefits to children at Odyssey Academy. The study will compare students' performance after intervention by comparing an intervention period to a standard care period, and comparing intervention students to students engaged in standard school activities in the area of academic performance.

DETAILED DESCRIPTION:
The objective of this study is to track if daily participation in motor lab activities for school age children improves their academic performance. Academic performance is associated with motor skills, coordination, and executive function. Our objectives are to determine if daily participation in motor lab activities changes these skills, to better understand these relationships, track outcomes of children participating in motor lab intervention compared to non-intervention and children receiving standard level of care in the school, and to be able to follow the intervention students over time.

The specific aims of the study are:

1. To investigate whether gross motor skills, fine motor skills, and physical fitness, predict executive function skills.
2. To determine the relationship between these variables and academic performance.
3. To examine the relationship between participation in motor lab activities and measures of change in fitness, gross motor skills, fine motor skills, executive function, and academic performance.
4. To evaluate if participation in daily motor lab activities predicts fitness level, gross motor skills, fine motor skills, executive function, and academic success at the end of the school year and in the next school year.

ELIGIBILITY:
Inclusion Criteria:

* students in grades kindergarten through fourth grade,
* students below grade level in reading
* in Odyssey Academy's reading program

Exclusion Criteria:

* students that are not part of the specialized reading program at Odyssey Academy
* are unwilling to participate in the motor lab intervention
* lack conversational ability in the use of the English language.

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Change in Movement Assessment Battery for Children-2 (MABC-2) between 3 time points (baseline, 10 weeks, 20 weeks) | Baseline, 10 weeks, 20 weeks
  Motor skills test which provides standard scores from 1-19 where higher scores represent better performance.
Change in Wechsler Intelligence Scale for Children-5 (WISC-5) between 3 time points (baseline, 10 weeks, 20 weeks) | Baseline, 10 weeks, 20 weeks
  Measures of executive function which provides scale scores from 1-19 where higher scores represent better performance.
Change in Test of Visual Motor Integration (VMI) between 3 time points (baseline, 10 weeks, 20 weeks) | Baseline, 10 weeks, 20 weeks
  Measures of visual perception and visual motor skills providing scores from 45-155 where higher scores represent better performance.
Change in Behavior Rating Inventory of Executive Function - Parent and Teacher Forms between 3 time points (baseline, 10 weeks, 20 weeks) | Baseline, 10 weeks, 20 weeks
  Measure of behavioral executive function with score within the range of 30-90 where scores >60 represent poorer performance.

SECONDARY OUTCOMES:
Change in Renaissance Star Reading Assessment between 3 time points (baseline, 10 weeks, 20 weeks) | Baseline, 10 weeks, 20 weeks
  Reading assessment with domain scores ranging from 0-99 where higher scores represent stronger performance.
Change in Fitness Gram between 3 time points (baseline, 10 weeks, 20 weeks) | Baseline, 10 weeks, 20 weeks
  fitness assessment with scores falling within either healthy fitness zone, needs improvement zone, or health risk zone.

IPD SHARING:
Plan to Share IPD: No